CLINICAL TRIAL: NCT02523833
Title: Evaluation of Small Airway Involvement in Patients With Chronic Hypersensitivity Pneumonitis and Its Impact on Exercise Limitation
Brief Title: Small Airway Involvement in Patients With Chronic Hypersensitivity Pneumonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Olívia Meira Dias, Medical doctor, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDC 3966/13/091
Record Dates: First submitted 2015-08-09; First posted 2015-08-14 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Hypersensitivity Pneumonitis; Airway Disease Small
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic HP patients (Other): Chronic hypersensitivity pneumonitis patients - use of salbutamol
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol — Salbutamol after spirometry, plethysmography and forced oscillation technique.
  Other Names: Aerolin

SUMMARY:
Hypersensitivity pneumonitis (HP) is a syndrome with variable clinical presentation in which lung inflammation is caused by inhalation of specific organic antigens or low molecular weight particles in previously sensitized individuals. Systemic symptoms may or may not be present. Chronic HP represents the final stage of the disease, caused by prolonged exposure to a particular antigen, leading to pulmonary fibrosis. In chronic HP, pulmonary function tests (PFTs) commonly present a restrictive ventilatory pattern, with decreased diffusion of carbon monoxide (DLCO). Some patients can also have obstructive disorders with expiratory flow limitation, due to obstruction of the small airways typically caused by bronchiolar involvement in this pathology. However, PFTs are relatively insensitive for detecting small airway involvement when there is concomitant interstitial fibrosis. First, conventional PFTs may be normal in patients with small airway involvement, since they contribute to less than 30% of the total airway resistance. In addition, damage to the small airways in HP is generally occurring parallel to areas of focal fibrosis - even when small airways are involved, these regions can be completely ignored, since they are excluded from ventilation. In summary, traditional PFTs are not sufficiently sensitive to detect diffuse small airway involvement in these diseases. In these cases, other functional tests, such as forced oscillation technique (FOT) and high resolution computer tomography (HRCT) scans of the chest with expired studies, could be used for this purpose.

This will be a cross-sectional study, which will include the following evaluations in 28 patients with HP recruited from our clinic:

- Clinical variables: (A) demographic and anthropometric data; (B) Clinical data: Onset of symptoms and time of diagnosis

C) Dyspnea score:

D) Smoking: * Current or former smoker * Smoking history (number of cigarettes smoked per day and for how long);

* Spirometry with forced and slow maneuvers before and after bronchodilator (salbutamol);
* Plethysmography to measure lung volumes;
* Diffusion capacity of carbon monoxide (DLCO);
* High-resolution chest CT with expiratory scans;
* Six-minute walk test;
* Cardio-respiratory test using a maximal incremental treadmill.
* Forced oscillation technique (FOT).

DETAILED DESCRIPTION:
Hypersensitivity pneumonitis (HP) is a syndrome with variable clinical presentation, in which inflammation in lung parenchyma is caused by inhalation of organic antigens or specific low molecular weight substances in previously sensitized individuals. Systemic symptoms may or not be present. Chronic HP represents the final stage of this disease, where prolonged exposure to a particular antigen would lead to lung fibrosis. The list of new antigens is growing, but the main antigens responsible for this disease are exposure to mold and birds.

Not all exposed individuals develop HP. The pathophysiology involves initial exposure and a subsequent decrease in antigen tolerance. Genetic susceptibility can also modulate the immune response to a specific antigen.

There are no reliable epidemiological data on the incidence or prevalence of HP. Differences in the type of antigen sensitization, lack of standardized diagnostic criteria and underreporting are possible factors. In Mexico, one of the few population surveys showed an estimated incidence of 30 cases per 100000 inhabitants in 2 years (1988-1990); however, there are some bias that limit the extrapolation of data to other contexts.

The patient rarely associates the onset of symptoms with a relevant exposure, making it important to actively search for environmental factors against respiratory complaints. It is believed that intermittent exposure to an antigen, long-term exposure to a small load of antigen or a cumulative effect of multiple episodes of acute exposure can cause chronic HP. It is noteworthy that only a small proportion of patients with a single episode of acute exposure will develop chronic HP.

In chronic HP, the patient complains of dyspnea on exertion and dry cough. Systemic symptoms such as fever and weight loss are rarely reported and may be associated with episodes of acute exposure. Physical examination reveals crackles and less commonly, digital clubbing. Auscultation may reveal the presence of squawks arising from the abrupt opening of small airways. Hypoxemia is found in patients with more severe lung disease.

The differential diagnosis with other fibrosing interstitial diseases is challenging, due to the overlap of clinical history, functional and tomographic findings in the terminal stages of these pathologies. There is no gold standard test for diagnosis of HP in all its forms: the diagnosis results in the combination of epidemiological, clinical, radiological data and other exams.

High resolution computer tomography (HRCT) has a fundamental role in the differential diagnosis. However, in advanced stages, the tomographic scans can demonstrate a pattern indistinguishable from nonspecific interstitial pneumonia (NSIP) or usual interstitial pneumonia (UIP), with presence of architectural distortion, traction bronchiectasis and bronchiolectasis, minimum ground glass opacities and honeycombing. The interpretation of HRCT allows "clues" for the differential diagnosis with other idiopathic intersticial pneumonias (IIPs). In comparative HRCT studies, there were some findings showing small airway involvement, such as lobular areas with decreased attenuation and vascularity, air trapping and ground glass or centrilobular micronodules Surgical biopsy may aid in the differential diagnosis of HP from other chronic idiopathic interstitial pneumonitis, especially when exposure is unclear. Even in advanced fibrosis, the accentuation of inflammation around the small airways is the major finding.

Pulmonary function tests (PFTs) commonly show restrictive ventilatory defect with decreased DLCO. There may be concomitant obstructive ventilatory defect, secondary to involvement of the small airways.

However, PFTs are relatively insensitive for detecting small airway involvement when there is concomitant interstitial fibrosis. Firstly, conventional PFTs may be normal in patients with involvement of small airways since they contribute to less than 30% of total airway resistance. Furthermore, damage to small airways in HP is generally focal occurring in parallel with fibrosed areas - even when small airways are involved, these regions may be completely disregarded since they are excluded from ventilation, with PFTs globally featuring a standard restrictive pattern.

In summary, traditional PFTs are not sensitive enough to detect diffuse small airway involvement in these diseases, no matter how severe it is, neither can detect focal changes. In these cases, the investigators hypothesize that other tests, such as forced oscillometry technique (FOT), with its experience widely recognized in the context of evaluation of obstructive diseases like asthma and chronic obstructive pulmonary disease (COPD) and the technique of negative expiratory pressure (NEP) could be used for this purpose. For now, imaging tests, especially high-resolution tomography with expiratory scans, seem to be more sensitive to detect small airway involvement.

Removal of the causal exposure is the treatment of choice. The use of corticosteroids reduces the duration of the acute phase, but does not affect long-term prognosis. Inhaled corticosteroids and bronchodilators may be used when there is evidence of airflow limitation, but there is no evidence basing its use.

2. Study hypothesis

The investigators' hypothesis is that a proportion of patients diagnosed with chronic HP exhibit expiratory flow limitation, due to airway obstruction caused mostly by the bronchiolar involvement characteristic of this pathology. This involvement could be quantified through other functional tests, such as FOT, and imaging techniques such as high resolution CT scan of the chest with expiratory scans. This may be one of the mechanisms that justifies the lower exercise capacity and greater degree of dyspnea on exertion in these individuals, together with other factors secondary to interstitial lung fibrosis, even in those patients with normal FEV1 (forced expiratory volume in 1 second) /FVC (forced vital capacity) , FEV1, residual volume (RV) and resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hypersensitivity pneumonitis confirmed by:

  * patients with known exposure to antigen, tomographic criteria and absence of other diagnoses;
  * confirmation with histology obtained by transthoracic biopsy, surgical biopsy or bronchoalveolar lavage with lymphocytosis above 30%;
* Age between 18 to 75 years;
* Clinically stable (no exacerbations or hospitalizations related to the underlying disease) for at least 6 weeks;
* Compliance with signing an informed consent for participation in the project.

Exclusion Criteria:

* Patients with FEV1 and / or DLCO <30% predicted;
* Patients using supplemental oxygen;
* Previous diagnosis of asthma or COPD;
* Pregnant women;
* Musculoskeletal disorders that limit exercise;
* Another medical condition that might interfere with the execution of tests;
* Current or past smoking history with tobacco intake greater than 30 pack-years;
* Severe heart disease functional class New York Heart Association (NYHA) III-IV) and / or decompensated hear failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Pletismography - forced expiratory volume in 1 second / forced vital capacity (FEV1/FVC) < 0.7, residual volume (VR) and VR/total lung capacity (TLC) values and changes with salbutamol | One day visit
  Percentage of VEF1/FVC < 0.7, residual volume (VR) >120% predicted and VR/total lung capacity (TLC)>.45 values and changes with salbutamol

SECONDARY OUTCOMES:
Air trapping in expiratory chest CT scans | One day visit
  Expiratory / inspiratory mean lung attenuation ratio as a measure of air trapping
Reactance and impedance of small airways through forced oscillation technique | One day visit
  Reactance and impedance of small airways

OTHER OUTCOMES:
Maximal cardiopulmonary exercise testing | One day visit
  Decrease of inspiratory capacity > 10% during maximal cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roberto R de Carvalho, MD, PhD, Principal Investigator — Heart Institute (InCor)
Locations (1):
- Olívia Meira Dias, São Paulo, Brazil

REFERENCES:
- [Background] Dellaca RL, Duffy N, Pompilio PP, Aliverti A, Koulouris NG, Pedotti A, Calverley PM. Expiratory flow limitation detected by forced oscillation and negative expiratory pressure. Eur Respir J. 2007 Feb;29(2):363-74. doi: 10.1183/09031936.00038006. Epub 2006 Nov 1. PMID 17079262
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Result] Lacasse Y, Selman M, Costabel U, Dalphin JC, Ando M, Morell F, Erkinjuntti-Pekkanen R, Muller N, Colby TV, Schuyler M, Cormier Y; HP Study Group. Clinical diagnosis of hypersensitivity pneumonitis. Am J Respir Crit Care Med. 2003 Oct 15;168(8):952-8. doi: 10.1164/rccm.200301-137OC. Epub 2003 Jul 3. PMID 12842854
- [Result] Selman M, Pardo A, Barrera L, Estrada A, Watson SR, Wilson K, Aziz N, Kaminski N, Zlotnik A. Gene expression profiles distinguish idiopathic pulmonary fibrosis from hypersensitivity pneumonitis. Am J Respir Crit Care Med. 2006 Jan 15;173(2):188-98. doi: 10.1164/rccm.200504-644OC. Epub 2005 Sep 15. PMID 16166619
- [Result] Lynch DA, Newell JD, Logan PM, King TE Jr, Muller NL. Can CT distinguish hypersensitivity pneumonitis from idiopathic pulmonary fibrosis? AJR Am J Roentgenol. 1995 Oct;165(4):807-11. doi: 10.2214/ajr.165.4.7676971.
- [Result] Silva CI, Muller NL, Lynch DA, Curran-Everett D, Brown KK, Lee KS, Chung MP, Churg A. Chronic hypersensitivity pneumonitis: differentiation from idiopathic pulmonary fibrosis and nonspecific interstitial pneumonia by using thin-section CT. Radiology. 2008 Jan;246(1):288-97. doi: 10.1148/radiol.2453061881. PMID 18096541
- [Result] Buschman DL, Gamsu G, Waldron JA Jr, Klein JS, King TE Jr. Chronic hypersensitivity pneumonitis: use of CT in diagnosis. AJR Am J Roentgenol. 1992 Nov;159(5):957-60. doi: 10.2214/ajr.159.5.1414806.